CLINICAL TRIAL: NCT00488111
Title: Fluid Management With Ringer's and 6% Starch for Cesarean Section After Epidural or Spinal Anesthesia
Brief Title: Fluid Management for Cesarean Section
Acronym: FMCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Maternal and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMU-2579FW; NMCH2007-221
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2008-08

CONDITIONS: Cesarean Section
Keywords: Regional anesthesia; Fluid Therapy; Hemostasis, Surgical
MeSH Terms: interventions — Ringer's Lactate; Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants were treated with normal Ringer's solution 15 min before the operation.
  Interventions: Other: Ringer's Lactate
- 2 (Active Comparator): 6% Starch was used 15min before operation followed epidural anesthesia.
  Interventions: Other: 6% Starch

INTERVENTIONS:
Other: Ringer's Lactate — Ringer's Lactate was used 15min before operation
  Other Names: RL
  Arms: 1
Other: 6% Starch — 6% Starch was used 15min before operation
  Other Names: ST
  Arms: 2

SUMMARY:
Cesarean section-associated hypotension is one of the pivotal factors to influence the Apgar Score of children and related with the stable hemostasis during the whole process of labor. How to keep circulation in a consistent stability is yet to be known. The investigators hypothesized that different fluids, crystalloids or colloids, can produced varying effects in keeping the physiological environment of labor from significant fluctuating.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 yr
* First time of delivery
* ASA status I-II
* No premature
* No genetic and infectious diseases
* Chinese

Exclusion Criteria:

* < 21 yr
* > 40 yr
* Subjects with cardiac and pulmonary disorders
* Dislocation of placenta
* Pregnant hypertension
* Allergy to local anesthetics
* Unwilling to cooperation
* Need intraoperative administration of vascular active agents
* With significant delivery side effects

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 850 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Total volume of colloid Total volume of crystalloid Total fluid volume | 6 months

SECONDARY OUTCOMES:
Percentage reduction in hematocrit, Days in hospital | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Care Hospital, Nanjing, Jiangsu, China